CLINICAL TRIAL: NCT00506675
Title: A Randomized Trial to Evaluate Combined Patching-Atropine for Residual Amblyopia
Brief Title: Combined Patching-Atropine for Residual Amblyopia
Acronym: ATS11
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment and infeasibility of ever reaching the necessary sample size
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-135; 2U10EY011751 (NIH)
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; Atropine; Patching
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive (Active Comparator): 42 hours per week of patching combined with atropine (1%) once daily in the sound eye, with spectacle correction (if needed)
  Interventions: Device: Patching; Drug: Atropine
- Weaning (Active Comparator): For patients currently patching, reduce patching to two hours daily for four weeks, then no treatment thereafter except spectacle correction (if needed). For patients currently using atropine, reduce atropine to once weekly for 4 weeks, then no treatment thereafter except spectacle correction (if needed)
  Interventions: Device: Patching; Drug: Atropine

INTERVENTIONS:
Device: Patching — 42 hours per week of patching
  Other Names: Coverlet, 3M Opticlude, Ortopad®
  Arms: Intensive
Drug: Atropine — daily atropine (1%)
  Arms: Intensive
Device: Patching — two hours of daily patching for 4 weeks, then no treatment
  Other Names: Coverlet, 3M Opticlude, Ortopad®
  Arms: Weaning
Drug: Atropine — once weekly atropine for 4 weeks, then no treatment
  Arms: Weaning

SUMMARY:
This study is designed to evaluate the effectiveness of treatment of residual amblyopia in children ages 3 to < 10 years with visual acuity of 20/32 to 20/63 in the amblyopic eye. The study is a randomized clinical trial comparing intensive treatment (42 hours per week of patching plus daily atropine) with a control group that will have rapid weaning of existing treatment followed by spectacle correction only (if needed). The primary objective is to determine if this intensive treatment will improve visual acuity in patients with residual amblyopia.

The primary outcome assessment is amblyopic eye visual acuity at 10 weeks.

The primary analytic approach for the amblyopic eye acuity will be a treatment group comparison of the proportion of patients with at least two lines of visual acuity improvement.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Both patching and atropine are accepted treatment modalities for the management of moderate amblyopia in children. Despite best efforts with conventional treatment, some patients fail to achieve normal visual acuity in the amblyopic eye. In a randomized trial conducted by PEDIG comparing atropine versus patching in 3 to 6 year olds with moderate amblyopia (ATS1), 261 of 402 patients (65%) had amblyopic eye visual acuity of 20/32 or worse after 6 months of treatment with patching or atropine. Beyond 6 months, treatment was at investigator discretion, and two years after randomization, 181 of 363 children (50%) still had amblyopic eye visual acuity of 20/32 or worse. In a randomized trial conducted by PEDIG comparing patching regimens, 129 of 181 patients with moderate amblyopia (71%) and 145 of 157 patients with severe amblyopia (92%) had amblyopic eye visual acuity of 20/32 or worse after 4 months of occlusion therapy. Many patients receive treatment beyond 6 months but still fail to achieve normal visual acuity in the amblyopic eye. It is unknown whether an intensive "final push" of combined treatment with daily patching and atropine will improve visual acuity in these patients. Although some clinicians prescribe simultaneous patching and atropine for selected patients, there are no published reports of its effectiveness. Also, we are not aware of reports of response to treatment of residual amblyopia.

The study has been designed as a simple trial that, other than the type of amblyopia therapy being determined through the randomization process, approximates standard clinical practice. Patients will be randomized to one of two treatment regimens:

* Intensive treatment: 42 hours per week of patching combined with daily atropine (1%)
* Control group: Weaning of the current treatment (two hours of daily patching for patients currently using patching and once weekly atropine for patients currently using atropine) for 4 weeks, then no treatment other than spectacles (if needed).

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to < 10 years
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye between 20/32 and 20/63 inclusive
* Visual acuity in the sound eye 20/32 or better and inter-eye acuity difference >= 2 logMAR lines
* Current/previous treatment with patching and/or atropine subject to the following stipulations:

  * No simultaneous treatment with patching and atropine in the past 6 months
  * No prior use of atropine in combination with the sound eye spectacle lens reduced by more than 1.50 D
  * Maximum level of any previous treatment:

    * Patching: up to 42 hours per week (averaging 6 hours daily)
    * Atropine: up to once daily
  * Current treatment with 42 hours per week patching or daily atropine
* No improvement in best-corrected amblyopic eye visual acuity between two consecutive visits at least 6 weeks apart using the same testing method and optimal spectacle correction (if needed), with no improvement defined as follows:

  * No lines of improvement
  * For patients tested using E-ETDRS, letter score that is no more than 4 letters improved
* Wearing spectacles with optimal correction (if applicable)
* Investigator ready to wean or stop treatment

Exclusion Criteria:

* Current vision therapy or orthoptics
* Ocular cause for reduced visual acuity
* Prior intraocular or refractive surgery
* Strabismus surgery planned within 10 weeks
* Known allergy to atropine or other cycloplegic drugs
* Known skin reactions to patch or bandage adhesives
* Down Syndrome present

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K. Wallace, M.D., Study Chair — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group (PEDIG) Writing Committee; Wallace DK, Kraker RT, Beck RW, Cotter SA, Davis PL, Holmes JM, Repka MX, Suh DW. Randomized trial to evaluate combined patching and atropine for residual amblyopia. Arch Ophthalmol. 2011 Jul;129(7):960-2. doi: 10.1001/archophthalmol.2011.174. No abstract available. PMID 21746992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2007 and March 2009, 27 subjects were randomized to the intensive group and 28 randomized to the weaning group.
Pre-assignment Details: Eligible subjects were aged 3-<10 with strabismic and/or anisometropic amblyopia, best-corrected amblyopic eye acuity of 20/32 to 20/63, interocular acuity difference greater than or equal to 2 lines, and no improvement in amblyopic eye acuity between 2 consecutive visits at least 6 weeks apart.
Groups:
- Intensive: 6 hours daily patching combined with daily atropine
- Weaning: For patients currently patching, a reduction of current treatment for 4 weeks with 2 hours daily patching or once weekly atropine followed by spectacles alone if needed.
Period: Overall Study
Arm/Group | Intensive | Weaning
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive | Weaning | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (1.1) | 6.9 (1.3) | 6.9 (1.2)
Age, Customized [Number; unit: participants] — Age at Enrollment in Years
  participants
    3 to < 7 years | 15 | 13 | 28
    7 to < 10 years | 12 | 15 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 13 | 17 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 22 | 40
  African American | 0 | 0 | 0
  Hispanic or Latino | 7 | 4 | 11
  Asian | 0 | 1 | 1
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55
Cause of Amblyopia [Number; unit: participants]
  Strabismus | 10 | 16 | 26
  Anisometropia | 6 | 3 | 9
  Strabismus and Anisometropia | 11 | 9 | 20
Current Treatment for Amblyopia at Enrollment [Number; unit: participants]
  Patching | 18 | 21 | 39
  Atropine | 9 | 7 | 16
Distance Visual Acuity in Amblyopic Eye [Number; unit: Participants] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  Participants
    20/63 (0.54 to 0.46 logMAR) | 3 | 2 | 5
    20/50 (0.44 to 0.36 logMAR) | 13 | 12 | 25
    20/40 (0.34 to 0.26 logMAR) | 7 | 10 | 17
    20/32 (0.24 to 0.16 logMAR) | 4 | 4 | 8
Distance Visual Acuity in Fellow Eye [Number; unit: Participants] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  Participants
    20/32 (0.24 to 0.16 logMAR) | 2 | 4 | 6
    20/25 (0.14 to 0.06 logMAR) | 10 | 7 | 17
    20/20 (0.04 to -0.04 logMAR) | 8 | 11 | 19
    20/16 (-0.06 to -0.14 logMAR) | 7 | 6 | 13
Refractive Error in Amblyopic Eye (spherical equivalent/diopters) [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  participants
    < 0.00D | 0 | 3 | 3
    0 to < +1.00 D | 1 | 0 | 1
    +1.00 to < +2.00D | 3 | 1 | 4
    +2.00 to < +3.00D | 0 | 2 | 2
    +3.00 to < +4.00D | 1 | 5 | 6
    greater than or equal to +4.00D | 22 | 17 | 39
Refractive Error in Fellow Eye [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  participants
    < 0.00D | 1 | 0 | 1
    0 to < +1.00D | 2 | 2 | 4
    +1.00 to < +2.00D | 5 | 5 | 10
    +2.00 to < +3.00D | 4 | 4 | 8
    +3.00 to < +4.00D | 6 | 7 | 13
    greater than or equal to +4.00D | 9 | 10 | 19
Mean (SD) Intereye Acuity Difference [Mean (Standard Deviation); unit: logMAR] — The difference between eyes in logMAR acuity was calculated with positive values indicating sound eye better. One letter = .02 logMAR, .1 logMAR = 5 letters or one line of visual acuity.
  logMAR | 0.33 (0.11) | 0.31 (0.10) | 0.32 (0.11)
Mean (SD) Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.02 (0.09) | 0.03 (0.10) | 0.03 (0.09)
Mean (SD) Spherical Equivalent Refractive Error in Amblyopic Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopters | 5.39 (2.33) | 4.24 (2.15) | 4.81 (2.29)
Mean (SD) Spherical Equivalent Refractive Error in Fellow Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopters | 3.46 (2.38) | 3.29 (1.90) | 3.37 (2.13)
Mean (SD) Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.35 (0.09) | 0.34 (0.08) | 0.35 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Amblyopic Eye Visual Acuity at 10 Weeks
Description: Visual acuity was measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 to 20/800 for ages 3 to <7; or with the electronic early treatment diabetic retinopathy study (E-ETDRS) method for 7 to <10 year olds which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
Time Frame: 10 Weeks
Measure: Number; unit: participants
Arm/Group | Intensive | Weaning
Number analyzed (Participants) | 27 | 28
participants
  20/125 (0.84 to 0.76 logMAR) | 0 | 1
  20/100 (0.74 to 0.66 logMAR) | 0 | 0
  20/80 (0.64 to 0.56 logMAR) | 1 | 1
  20/63 (0.54 to 0.46 logMAR) | 1 | 4
  20/50 (0.44 to 0.36 logMAR) | 4 | 0
  20/40 (0.34 to 0.26 logMAR) | 13 | 9
  20/32 (0.24 to 0.16 logMAR) | 7 | 7
  20/25 (0.14 to 0.06 logMAR) | 1 | 3
  20/20 (0.04 to -0.04 logMAR) | 0 | 2
  20/16 (-0.16 to -0.24 logMAR) | 0 | 0
Statistical Analysis 1: Comparison: Intensive vs Weaning; Test type: Superiority or Other; p = 0.30, ANCOVA

2. Primary Outcome: Mean (SD) Distribution of Visual Acuity at 10 Weeks
Description: as for outcome 1
Time Frame: 10 Weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Intensive | Weaning
Number analyzed (Participants) | 27 | 28
logMAR | 0.30 (0.10) | 0.29 (0.18)
Statistical Analysis 1: Comparison: Intensive vs Weaning; Test type: Superiority or Other; p = 0.30, ANCOVA

3. Primary Outcome: Distribution of Amblyopic Eye Visual Acuity Change From Baseline to 10 Weeks
Description: Change in logMAR from baseline to 10 weeks was calculated, with positive difference indicating improvement. Note one logMAR line = 5 letters or one Snellen line equivalent.
Time Frame: baseline to 10 Weeks
Measure: Number; unit: Participants
Arm/Group | Intensive | Weaning
Number analyzed (Participants) | 27 | 28
Participants
  greater than or equal to 3 lines | 0 | 1
  2 to < 3 lines worse | 1 | 0
  1 to < 2 lines worse | 2 | 4
  Within 1 logMAR line | 12 | 8
  1 to < 2 lines better | 9 | 8
  2 to < 3 lines better | 3 | 5
  greater than or equal to 3 lines better | 0 | 1
Statistical Analysis 1: Comparison: Intensive vs Weaning; Test type: Superiority or Other; p = 0.30, ANCOVA

4. Primary Outcome: Mean (SD) Change in Visual Acuity in the Amblyopic Eye at the 10 Week Primary Outcome Exam
Description: as for outcome 3
Time Frame: baseline to 10 Weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Intensive | Weaning
Number analyzed (Participants) | 27 | 28
logMAR | 0.056 (0.096) | 0.053 (0.150)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Intensive | Weaning
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 6/27 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=27) | Weaning (N=28)
Light sensitivity (General disorders) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was stopped after 18 months due to inadequate recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No